CLINICAL TRIAL: NCT02911168
Title: A Prospective, Randomized Comparison Between the Ultrasound Guided Paravertebral Block and the Ultrasound Guided Proximal Intercostal Nerve Block
Brief Title: Comparison of US-Guided Paravertebral and Proximal Intercostal Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kamen Vlassakov, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2016P000174/MGH
Record Dates: First submitted 2016-08-12; First posted 2016-09-22 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pain
Keywords: NERVE BLOCK; ANESTHESIA RECOVERY PERIOD; PAIN MANAGEMENT
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proximal Intercostal Block (Active Comparator): See Intervention Section
  Interventions: Procedure: Proximal Intercostal Block
- Paravertebral Block (Active Comparator): See Intervention Section
  Interventions: Procedure: Paravertebral Block

INTERVENTIONS:
Procedure: Proximal Intercostal Block — After identifying the correct intercostal space, the ultrasound probe will be moved medially to identify the transverse processes, then again laterally from the transverse processes to rest over the ribs so as to obtain the best view of ribs and pleura. A 10cm, 21G needle will be inserted in-plane at the caudal border of the probe. An attempt will be made to keep the needle tip and the target injection position (just under the internal intercostal membrane (IIM)) in view. Correct needle tip placement will be demonstrated by depression of the pleura/endothoracic fascia upon local anesthetic injection and by lack of retrograde spread of LA over the muscles or the ribs. The LA will be injected in 4 cc aliquots after negative aspiration of air, CSF and blood.
  Other Names: PICB
  Arms: Proximal Intercostal Block
Procedure: Paravertebral Block — After identifying the correct intercostal space, the ultrasound probe will be placed between the adjacent transverse processes in a longitudinal/parasagittal plane measuring 2.5cm from the midline. The best possible view of the transverse processes, the superior costotransverse ligament and pleura will be obtained. An attempt will be made to keep the needle tip and the target injection position (immediately beneath the costotransverse ligament) in view. Correct placement of the needle tip will be demonstrated by depression of the pleura upon injection of local anesthetic and by lack of retrograde spread of LA over the muscles or transverse processes. The LA will be injected in 4 cc aliquots after confirming negative aspiration of air, CSF and blood.
  Other Names: PVB
  Arms: Paravertebral Block

SUMMARY:
The purpose of this study is to compare the proximal intercostal block to the more medial (classic) ultrasound-guided paravertebral block. The investigators hypothesize that the proximal intercostal block will allow for improved needle visualization, shorter block time, and improved safety profile compared to the classic paravertebral bock.

DETAILED DESCRIPTION:
Although previous studies have made advances towards applying ultrasound guidance to the performance of paravertebral blocks (PVB), a technique combining both safety and technical ease remains elusive. The ideal technique (1) permits continuous visualization of the entire needle shaft and tip, (2) avoids aiming the needle tip and injectate directly toward the neuraxis or lung, and (3) is easy to perform. Visualization of all structures by ultrasound is essential to minimize the risk of vascular puncture, nerve root or spinal cord injury, and pneumothorax. Failure to consistently and quickly identify the transverse process and pleura, as occurs when using older techniques, results in several needle redirections, causing pain and discomfort to patients, and increases the potential risk of pneumothorax. The technical difficulty of applying previously-described US-guided techniques takes an inordinate amount of time and is clinically less practical within a busy surgical practice.

In the current study, the investigators describe a novel, modified approach to real-time ultrasound-guided single shot paravertebral blockade, the proximal intercostal block (PICB), which utilizes a sagittal paramedian US probe placement to identify the intercostal space and PVS. In this method, instead of placing the probe at a fixed traditional distance of 2.5 cm from the spinous processes, the probe is moved laterally to obtain a comprehensive image, with a clear view of the ribs, internal intercostal membrane, and the parietal pleura.

The investigators propose that moving the probe laterally towards the proximal intercostal space allows clearer simultaneous visualization of both pleura and needle as it advances towards the PVS, while achieving comparable injectate spread and, ultimately, similar or better clinical results. Such improved visualization will reduce the number of needle passes, increase confidence in the user, decrease block placement time, and improve overall block success. This technique combines the advantages of more lateral approaches (better visualization of structures, in particular the pleura) with the advantage of the more medial approaches (in-plane, closer, and not directed at the neuraxis).

ELIGIBILITY:
Inclusion Criteria:

1. Females age 18-85 years old
2. ASA 1-3
3. Patient scheduled for unilateral or bilateral mastectomy with or without reconstruction

Exclusion Criteria:

1. Coagulopathy
2. Patient refusal
3. Allergy to local anesthetics

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Ultrasound Image Quality Score | Evaluated at time of block
  The following will be assessed for each image and video, and saved during each block performed:
  1. Best possible image of block anatomy (including the pleura, transverse process/rib, costotransverse ligament/internal intercostal membrane, as appropriate) as well as needle location.
  2. Video of the space during injection, reflecting the injectate spread. The images will be rated by a separate regional anesthesiologist not involved in study, but proficient with both types of blocks and ultrasound imaging.
  3. The following score 3 point scale will be used to rate visibility: 0=not visible, 1=hardly visible, 2=well visible, 3=very well visible. Maximum score possible=18 including both pieces of media.

SECONDARY OUTCOMES:
Block Performance Time | Evaluated at time of block
  Defined as the sum of imaging and needling times
Imaging Time | Established during block performance
  Defined as the time interval between contact of the ultrasound probe with the patient, and the acquisition of a satisfactory image (which will be saved and analyzed later by a regional anesthesiologist blinded to the particular aims of the study).
Needling Time | Established during block performance
  Defined as the time interval between the start of the skin wheal and the end of local anesthetic injection through the block needle.
Number of Needle Passes | Established during block performance
  Initial needle insertion will be counted as "first pass". Any subsequent needle advancement, preceded by a retraction of more than 2 cm, will be counted as an additional pass.
Distance of Injection Sites from Midline | Established during block performance
  Measured and recorded (one of our clinical aims)
Presence of Perioperative Block-Related Complications | Within 24 hours of block placement
  The presence of the following complications will be recorded:
  1. Horner's syndrome
  2. Pneumothorax
  3. Local anesthetic systemic toxicity (LAST)
  4. Pain on injection
  5. Evidence of contralateral block (for unilateral procedures)
Effectiveness of the Block | One hour following extubation, and at 24 hours following block placement
  Patients will be asked to provide a verbal rating score of pain (0-10) at two time points: one hour following extubation, and 24h following block placement. At the 1 hour following extubation time point, we will be checking the coverage of the block in terms of dermatomal spread (see below).
Dermatomal spread | One hour following extubation
  Number of dermatomal block levels, determined by loss of sensation to cold (ice) or to loss of pinprick sensation in the PACU one hour after extubation.
Opioid requirement | Evaluated at 1 hour after extubation, and then at 24 hours following the block
  Opioid requirement, including intraoperative, PACU, and during the entire hospital admission, normalized to morphine equivalents.
Prolonged postoperative pain | 6 and 12 months after surgery
  Postoperative contact via secure e-mail at will assess for the incidence of chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kamen Vlassakov, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Fleischmann K. Ultrasound-guided thoracic parvertebral blocks: anatomy , approaches and techniques. Asra. 2012.
- [Background] Luyet C, Herrmann G, Ross S, Vogt A, Greif R, Moriggl B, Eichenberger U. Ultrasound-guided thoracic paravertebral puncture and placement of catheters in human cadavers: where do catheters go? Br J Anaesth. 2011 Feb;106(2):246-54. doi: 10.1093/bja/aeq309. Epub 2010 Nov 25. PMID 21112880
- [Background] Eason MJ, Wyatt R. Paravertebral thoracic block-a reappraisal. Anaesthesia. 1979 Jul-Aug;34(7):638-42. doi: 10.1111/j.1365-2044.1979.tb06363.x. PMID 517716
- [Background] Naja Z, Lonnqvist PA. Somatic paravertebral nerve blockade. Incidence of failed block and complications. Anaesthesia. 2001 Dec;56(12):1184-8. doi: 10.1046/j.1365-2044.2001.02084-2.x. PMID 11736777
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876
- [Background] Naja MZ, Ziade MF, Lonnqvist PA. Nerve-stimulator guided paravertebral blockade vs. general anaesthesia for breast surgery: a prospective randomized trial. Eur J Anaesthesiol. 2003 Nov;20(11):897-903. doi: 10.1017/s0265021503001443. PMID 14649342
- [Background] Mehta Y, Arora D, Sharma KK, Mishra Y, Wasir H, Trehan N. Comparison of continuous thoracic epidural and paravertebral block for postoperative analgesia after robotic-assisted coronary artery bypass surgery. Ann Card Anaesth. 2008 Jul-Dec;11(2):91-6. doi: 10.4103/0971-9784.41576. PMID 18603748
- [Background] Richardson J, Cheema SP, Hawkins J, Sabanathan S. Thoracic paravertebral space location. A new method using pressure measurement. Anaesthesia. 1996 Feb;51(2):137-9. doi: 10.1111/j.1365-2044.1996.tb07700.x. PMID 8779368
- [Background] Pusch F, Wildling E, Klimscha W, Weinstabl C. Sonographic measurement of needle insertion depth in paravertebral blocks in women. Br J Anaesth. 2000 Dec;85(6):841-3. doi: 10.1093/bja/85.6.841. PMID 11732516
- [Background] O Riain SC, Donnell BO, Cuffe T, Harmon DC, Fraher JP, Shorten G. Thoracic paravertebral block using real-time ultrasound guidance. Anesth Analg. 2010 Jan 1;110(1):248-51. doi: 10.1213/ANE.0b013e3181c35906. Epub 2009 Nov 21. PMID 19933536
- [Background] Ben-Ari A, Moreno M, Chelly JE, Bigeleisen PE. Ultrasound-guided paravertebral block using an intercostal approach. Anesth Analg. 2009 Nov;109(5):1691-4. doi: 10.1213/ANE.0b013e3181b72d50. PMID 19843811
- [Background] Burns DA, Ben-David B, Chelly JE, Greensmith JE. Intercostally placed paravertebral catheterization: an alternative approach to continuous paravertebral blockade. Anesth Analg. 2008 Jul;107(1):339-41. doi: 10.1213/ane.0b013e318174df1d. PMID 18635506
- [Background] Renes SH, Bruhn J, Gielen MJ, Scheffer GJ, van Geffen GJ. In-plane ultrasound-guided thoracic paravertebral block: a preliminary report of 36 cases with radiologic confirmation of catheter position. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):212-6. doi: 10.1097/aap.0b013e3181c75a8b. PMID 20301827
- [Background] Marhofer P, Kettner SC, Hajbok L, Dubsky P, Fleischmann E. Lateral ultrasound-guided paravertebral blockade: an anatomical-based description of a new technique. Br J Anaesth. 2010 Oct;105(4):526-32. doi: 10.1093/bja/aeq206. Epub 2010 Aug 3. PMID 20685684
- [Background] Abdallah FW, Brull R. Off side! A simple modification to the parasagittal in-plane approach for paravertebral block. Reg Anesth Pain Med. 2014 May-Jun;39(3):240-2. doi: 10.1097/AAP.0000000000000086. PMID 24682082
- [Background] Karmakar MK, Li X, Kwok WH, Ho AM, Ngan Kee WD. Sonoanatomy relevant for ultrasound-guided central neuraxial blocks via the paramedian approach in the lumbar region. Br J Radiol. 2012 Jul;85(1015):e262-9. doi: 10.1259/bjr/93508121. Epub 2011 Oct 18. PMID 22010025
- [Derived] Vlassakov K, Vafai A, Ende D, Patton ME, Kapoor S, Chowdhury A, Macias A, Zeballos J, Janfaza DR, Pentakota S, Schreiber KL. A prospective, randomized comparison of ultrasonographic visualization of proximal intercostal block vs paravertebral block. BMC Anesthesiol. 2020 Jan 9;20(1):13. doi: 10.1186/s12871-020-0929-x. PMID 31918668